CLINICAL TRIAL: NCT03251937
Title: VERITAS - A Study to Demonstrate the Value of Multiple Modalities Using the Spectra WaveWriter™ Spinal Cord Stimulator System in the Treatment of Chronic Pain
Brief Title: Value of Multiple Modalities Using the Spectra WaveWriter Spinal Cord Stimulator System
Acronym: VERITAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A4064
Record Dates: First submitted 2017-08-15; First posted 2017-08-16 (Actual); Results first posted 2020-03-16 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Chronic Pain; Back Pain
Keywords: Chronic Pain; Back Pain; Leg Pain; Pain; Stimulation; Spinal Cord Stimulator; Implantable Pulse Generator
MeSH Terms: conditions — Chronic Pain; Back Pain; Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Spinal Cord Stimulation (Experimental): Spectra WaveWriter SCS System
  Interventions: Device: Spectra WaveWriter SCS System

INTERVENTIONS:
Device: Spectra WaveWriter SCS System — Multiple modalities of stimulation therapy
  Other Names: Spectra WaveWriter Spinal Cord Stimulation System

SUMMARY:
To demonstrate the value of multiple modalities and sustained clinically significant pain relief in patients with chronic pain when using the Boston Scientific Spectra WaveWriter Spinal Cord Stimulator (SCS) System.

ELIGIBILITY:
Key Inclusion Criteria:

* Chronic pain of the trunk and/or limbs
* 22 years of age or older at time of enrollment
* Willing and able to comply with all protocol-required procedures and assessments/evaluations provided in English
* Willing and capable of giving informed consent

Key Exclusion Criteria:

* Any pain-related diagnosis or medical/psychological condition that, in the clinician's best judgment, might confound reporting of study outcomes
* Significant cognitive impairment that, in the opinion of the Investigator, would reasonably be expected to impair the study candidate's ability to participate in the study
* Current systemic infection, or local infection in close proximity to the anticipated surgical field
* Breast-feeding, pregnant or planning to get pregnant during the course of the study or not using adequate contraception
* Previous spinal cord stimulation trial or is already implanted with an active implantable device(s) (e.g. pacemaker, drug pump, implantable pulse generator)
* Participating, or intends to participate, in another clinical trial that may influence the data that will be collected for this study

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2018-01-09 (Actual); Primary Completion 2019-01-09 (Actual); Study Completion 2020-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roshini Jain, Study Director — Boston Scientific Corporation
Locations (15):
- United States (15):
  - Neurovations, Napa, California
  - Louis J. Raso, MD, PA, Jupiter, Florida
  - Florida Pain Clinic, Ocala, Florida
  - Forest Health Medical Center, Ypsilanti, Michigan
  - Mercy Medical Research Institute, Springfield, Missouri
  - University of Rochester, Rochester, New York
  - The Center for Clinical Research, LLC, Winston-Salem, North Carolina
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Western Reserve Spine and Pain Institute, Kent, Ohio
  - Toledo Clinic, Toledo, Ohio
  - West Chester Hospital, LLC, West Chester, Ohio
  - Pacific Sports and Spine, LLC, Eugene, Oregon
  - Spine Team Texas, Rockwall, Texas
  - Swedish Neuroscience Institute, Seattle, Washington
  - Advanced Pain Management Appleton, Appleton, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were considered enrolled once informed consent was completed. Only those who met all eligibility criteria went on to receive implant and proceed in the study.
Period: Overall Study
Arm/Group | Spinal Cord Stimulation
Started | 40
Completed | 37
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Spinal Cord Stimulation
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.2 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 40

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With 50% or Greater Reduction in Overall Pain From Baseline
Time Frame: 3 months post activation
Measure: Count of Participants; unit: Participants
Arm/Group | Spinal Cord Stimulation
Number analyzed (Participants) | 40
Participants | 31

ADVERSE EVENTS:
Time Frame: Adverse Events were collected through the entire study (up to 1 year post-activation) for all enrolled subjects in the study
Description: Adverse Events were collected through the entire study (up to 1 year post-activation) for all enrolled subjects in the study
Arm/Group | Spinal Cord Stimulation
All-Cause Mortality (participants affected / at risk) | 1/97
Serious Adverse Events (participants affected / at risk) | 7/97
Other Adverse Events (participants affected / at risk) | 0/97
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Spinal Cord Stimulation (N=97)
Angina (Cardiac disorders) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 1 (1)
Sinus Node Dysfunction (Cardiac disorders) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1)
Cerebrovascular Accident (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-10): https://cdn.clinicaltrials.gov/large-docs/37/NCT03251937/Prot_SAP_001.pdf